CLINICAL TRIAL: NCT03968380
Title: Contextualizing Evidence for Action on Diabetes in Low-resource Settings: a Mixed-methods Case Study in Quito and Esmeraldas, Ecuador.
Brief Title: Contextualizing Evidence for Action on Diabetes - Population Survey
Acronym: CEAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Lucy Anne Parker, Lecturer, Universidad Miguel Hernandez de Elche
Other Study IDs: ERC-2018-STG-804761
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Implementation science; Noncommunicable disease; Diabetes Mellitus, Type 2; Public Policy; Delivery of Health Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Noncommunicable Diseases | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population in Quito: 720 randomly chosen people living in District 17D06, Quito (Ecuador)
  Interventions: Other: Population survey with biological and physical measurements.
- Population in Esmeraldas: 720 randomly chosen people living in Eloy Alfaro District, Esmeraldas (Ecuador)
  Interventions: Other: Population survey with biological and physical measurements.

INTERVENTIONS:
Other: Population survey with biological and physical measurements. — Individuals will be interviewed in their homes by trained interviewers. At a later date, in a location agreed with the study team, a sample of blood will be taken and we will measure fasting glucose, cholesterol level and creatinine. We will measure participants' height, weight, waist circumference and blood pressure. An Oral Glucose Tolerance Test (OGTT) will be performed on non-diabetic and/or non-pregnant participants.

SUMMARY:
This protocol reflects the first part of a larger mixed-methods study aimed at exploring the process by which global recommendations can be translated into context-specific, evidence-informed action for diabetes prevention in low-resource settings. The CEAD project will be carried out in 2 low-resource settings in Ecuador. Here, in recognition that rigorous epidemiological data on diabetes risk and morbidity is needed to explore applicability of potential actions, the investigators will undertake 2 representative cross-sectional population survey using geospatial sampling. We will collect dat by interview in the homes of the participants using WHO STEPS questionnaires and measure participants' physical and biological parameters.

DETAILED DESCRIPTION:
Objective: To provide rigorous epidemiological data on diabetes risk and morbidity in Health District 17D06 in Quito, Ecuador; and Eloy Alfaro District, located in the coastal region of Esmeraldas.

Design: The investigators will undertake two cross-sectional population surveys, with representative samples of the selected health districts, to estimate the prevalence of diabetes, impaired glucose tolerance, and NCD risk factors.

Sample design: Participants will be selected using multi-stage cluster sampling. We will use parishes or 'micro-areas' as primary Enumeration Areas (EA) for which official GIS shape files and population estimates are available. The EAs will be randomly selected with a probability proportional to its population density. In urban areas, after having sampled EAs, buildings or homes will be identified by randomly generated GPS points. The investigators will then sample one person at random in each household.

In rural areas, the investigators will randomly select villages from within the samples EAS, and then undertake the simple random sampling of individuals by using an existing census already developed by voluntary health promotors, and digitised by a local NGO. This census will be updated in the 3 months preceding sample selection to ensure accuracy.

Sample size: The sample size is proposed assuming the prevalence of diabetes is no higher than 10%, to provide an estimate with an absolute precision of +/- 3%, with a 95% confidence level. The investigators assume a design effect of 1.5 (recommended in STEPS guideline for complex designs in absence of locally available alternatives) and will further increased the sample size to allow for up to 20% refusal or loss due to individuals not attending their appointment for physical and biological measurements.

Survey procedures: The questionnaire will be designed according to the WHO STEPS NCD risk factor survey forms , and some survey-specific questions. Detailed demographic information will also be included following the WHO STEPS core questions and extended questions (highest level of education, ethnicity, marital status, employment status and household income). Cultural adaptations to the questions will be made as required.

The questions will be used to compile a purpose designed electronic survey form loaded onto tablets purchased for the research. The survey tool will be pre-piloted before the survey, after training the data collection team.

Thirty trained interviewers will establish survey eligibility, solicit informed consent, and carry out the survey in the participant's home. Composition of the survey team will be gender balanced, and include staff who represent local cultural, ethnic and religious groups. The survey will be carried out in Spanish but some interviewers will also be fluent in Quechua, Chachi and any other relevant indigenous language to translate questions verbally if required. Data collection in rural areas will engage the volunteer health promotors. The surveyors will arrange an appointment for physical and biological measurements together with the participant considering geographical convenience and availability. Individuals with a fasting blood glucose ≥ 126 mg/dl and/or a 2 hour plasma glucose ≥ 200 mg/dl, or blood pressure over 140/90 mmHg will be referred to their local health facility for care. All participants will receive the results of their physical measurements and blood analyses and will receive a health promotion booklet about diabetes, cardiovascular risk, and the importance of healthy diet and physical activity.

Physical measurements and laboratory: Weight, height, waist circumference will be measured and we will include limited biochemical measurements (fasting blood glucose, cholesterol and creatinine) analysed at regional reference laboratories. Participants will also undergo an Oral Glucose Tolerance Test (OGTT). Survey participants will be invited to a well-lit hygienic location after at least 8 hours fasting. Appointments will be first thing in the morning and participants will be instructed to eat or drink nothing but water from 10pm the night before. Instructions for fasting will be given on the appointment card given to the participants the survey day and telephone reminders will be sent when possible. All participants will receive breakfast after the OGTT test. Diabetic patients on medication will be asked to bring their medication and take it immediately after their breakfast after blood draw. They will not be asked to complete an OGTT. Similarly, pregnant women are eligible to participate in the study but will not undergo an OGTT, only fasting blood glucose. In order to ensure absence of pregnancy, the investigators will provide pregnancy tests to women in fertile age who are unable to confirm the absence of pregnancy at the household interview. Steps will be taken to minimise variability (at study zone level) in the pre-analytical treatment of samples. Blood extraction, storage and transportation will follow standard infection control measures.

Data management and analysis: Stickers with Quick Response (QR) codes that can be scanned by the android devices at each step will be used to ensure linkage of data collected in participant's home, their physical and biological measurements and laboratory results. The investigators will use and modify the WHO STEPS forms where possible and import them to Kobo toolbox free open source software (or ODK collect if necessary). Stata/SE (StataCorp, Texas, U.S.A.) Version 12.1. will be used for statistical analysis. The prevalence of impaired glucose tolerance, diabetes, and the other NCD risk factors will be calculated with 95% confidence intervals. Outcomes will be disaggregated by sex, age group, ethnicity and socioeconomic position. Geographical variation in survey outcomes will also be described. Steps will be taken to prevent missing data, but some level is unavoidable and we will incorporate methods analysing missing data or data from uncertain sources when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Providing written informed consent
* Current residence in the study area, defined as at least 20 days of the previous month sleeping in a residence in study zone and no plan to move in the foreseeable future.

Exclusion Criteria:

* Unability to provide informed consent (e.g. significant mental impairment)
* Pregnant women and diabetic patients will be excluded from participation on the oral glucose tolerance test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Geospatial sampling to achieve a representative sample of people aged 18 or more who are currently living in District 17D06, Quito, or Eloy Alfaro District, Esmeraldas (Ecuador), and are able to provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Glucose Tolerance | Blood sampling 2 hours after drinking a glucose solution of known concentration
  New cases of diabetes will be identified by performing the Oral Glucose Tolerance Test. Participants will drink a solution containing 75 g of glucose and their plasma glucose will be measured 2 hours later. Glucose concentration will be given in mg/dl. Individuals will be classified as having impaired glucose tolerance if glycemia after 2 hours is higher than 200 mg/dl and at risk of developing diabetes if he or she has a glicaemia between 140 and 199 mg/dl. Already diagnosed diabetic patients and pregnant women will not undergo this test.

SECONDARY OUTCOMES:
Fasting blood glucose | Venous blood sampling will be the first thing in the morning after at lease 8 hours fasting.
  We will measure fasting blood glucose using venous blood samples analysed at regional reference laboratories. Results will be given in mg/dl and we will consider an individual to have impaired fasting blood glucose if their value is higher than 126 mg/dl.
Obesity | At the moment of the survey
  Obesity will be measured as a body mass index equal or higher to 30, being body mass index defined as weight divided by squared height. Weight will be measured in kg and height in cm.
  Weight, height, and waist circumference will be measured in according to the technical specifications recommended in the STEPS guideline, in a separate area to ensure participant privacy.
Blood pressure | At the moment of the survey
  We will measure participants' blood pressure in a separate room ensuring privacy. Measurements will be taken twice within a 2-minute interval to ensure reliability. If values differ more than 5 mmHg, a third measurement will be taken and the final value will be the average of the three measured pressures. Results will be given in mmHg and we will consider an individual to have arterial hypertension if their blood pressure exceeds 90/140 mmHg for diastolic and systolic pressure, respectively.
Cholesterol | Venous blood sampling will be the first thing in the morning after at least 8 hours fasting.
  We will measure blood cholesterol using venous blood samples analysed at regional reference laboratories. Results will be given in mg/dl and we will consider an individual to have high blood cholesterol if their value is higher than 200 mg/dl.
Tobacco consumption | At time of survey, or ever. Frequency for current smokers measured with reference to usual days and weeks.
  We will ask participants about their tobacco consumption including frequency and type of products (number of cigarettes, cigars, etc per day or week) as well as past habits, starting age and whether they have tried to quit smoking.
  The questionnaire used for this purpose will include sections of the WHO STEPS NCD risk factor survey forms and cultural adaptations will be made as required.
Alcohol consumption | At time of survey, in reference to the previous week, month and over the 12 months prior to survey.
  We will ask participants about their current and past drinking habits including type of drink and monthly, weekly or daily frequency.
  The questionnaire used for this purpose will include sections of the WHO STEPS NCD risk factor survey forms and cultural adaptations will be made as required.
Fruit and vegetable intake | At time of survey in reference to usual days and weeks.
  We will ask participants about their weekly consumption of fruit and vegetables. The questionnaire used for this purpose will include sections of the WHO STEPS NCD risk factor survey forms and cultural adaptations will be made as required.
Physical activity | At time of survey in reference to usual days and weeks.
  We will ask participants about their physical activity patterns. We will include questions addressing moderate or vigorous physical activity as part of their work, traveling habits (walking, bicycle) or whether they practice any sport or physical exercise as a recreational activity.
  The questionnaire used for this purpose will include sections of the WHO STEPS NCD risk factor survey forms and cultural adaptations will be made as required.
Waist circumference | At time of survey.
  Waist circumference will be measured in cm and we will consider an individual to have high cardiovascular risk if it is higher than 88 cm for women and 102 cm for men.
  Weight, height, and waist circumference will be measured in according to the technical specifications recommended in the STEPS guideline, in a separate area to ensure participant privacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Mari Carmen Bernal Soriano, Esmeraldas, Ecuador